CLINICAL TRIAL: NCT03853356
Title: Evidence For Fusion In Spine With Orthoss®
Acronym: EFFISO
Status: Active, not recruiting | Type: Observational
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 13570-222
Record Dates: First submitted 2019-02-11; First posted 2019-02-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Spondylolisthesis Involving L4-L5; Lumbar Spondylolisthesis Involving L5-S1; Lumbar Spinal Stenosis; Lumbar Disc Degeneration
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lumbar spondylodesis involving 1-2 levels (L4-L5 and/or L5-S1): All surgical procedures to be performed during this clinical trial are part of the routine procedures for lumbar spondylodesis by using transforaminal lumbar interbody fusion (TLIF) and posterior lumbar interbody fusion (PLIF) techniques in the 1-2 levels (L4-L5 and/or L5-S1). Patients will receive surgery according to standard procedures.
  Interventions: Device: Orthoss

INTERVENTIONS:
Device: Orthoss — Orthoss® granules. Orthoss® granules mixed with local bone and pedicle bone marrow aspirate.

SUMMARY:
This study aims to evaluate the performance and safety of the Orthoss® as a bone graft extender in lumbar spondylodesis involving 1-2 levels (L4-L5 and/or L5-S1).

DETAILED DESCRIPTION:
This clinical investigation is a prospective, non-interventional, uncontrolled clinical trial, organized to generate clinical data on performance and safety of Orthoss® as a bone graft extender mixed with local bone at ratio of 1:1 and pedicle bone marrow aspirate in lumbar spondylodesis involving 1-2 levels. (Orthoss® is CE marked for this indication).

If you as a patient have a wear and tear disease of the spine, an operation serves to restore the stability of the spinal column. In order to promote a bony build-up of the lumbar spine segment (fusion), bone replacement material is used in your case as standard. The aim of this observational study is to determine fusion in order to address clinical performance of that bone replacement material.

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or female) must be 18 years or older
* The patient must be a candidate diagnosed with either degenerative disc disease including 1-2 level (L4-L5 and/or L5-S1) or dysplasic spondylolisthesis (degree 1 or 2) or lumbar stenosis
* If the patient is of child-bearing potential, the patient confirms not to be pregnant
* The patient is able to comply with the clinical investigation-related procedures such as attending all follow-up procedures
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent including the use of the anonymized data for scientific publication
* The patient will not participate in another clinical investigation during this clinical investigation

Exclusion Criteria:

* General contraindications for surgical treatment are present
* The patient has a history of malignancy, radiotherapy, or chemotherapy for malignancy within the past five years
* The patient is currently being treated with radiation, chemotherapy, immunosuppression or steroid therapy dose equivalent of more than 5mg prednisolon
* The patient is pregnant or nursing
* Women of childbearing age who are not using a highly effective method of birth control
* The patient has acute or chronic infection at the surgical site
* The patient has a known allergy to bovine bone material
* The patient has a medical history of alcohol or drug abuse within the last year prior to the screening examination
* Vulnerable population
* Patient is currently participating, or has participated in another clinical investigation within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Orthoss® mixed with local bone and pedicle bone marrow aspirate in lumbar spondylodesis by using transforaminal lumbar interbody fusion (TLIF) and posterior lumbar interbody fusion (PLIF) techniques in the 1-2 levels.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | 6 months
  Successful fusion should be based on the translational motion < 3mm as well as on the angular motion < 5° at 6 months.

SECONDARY OUTCOMES:
Clinical Outcome Measure - Quality of Life: Oswestry Low Back Disability Index | 1-4 weeks; 3, 6, 12 and 24 months
  Improvement in Oswestry Low Back Disability Index (ODI) of 15 or more at 24 months from the pre-operative value.Zero is equated with no disability and 100 is the maximum disability possible.
Clinical Outcome Measure - Leg pain | 1-4 weeks, 3,6,12 and 24 months
  Decrease in Visual Analog Scale for Pain (VAS) for leg by 3/10 or more at 24 months from the pre-operative value. Patients rated their leg pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score fo 10 representing "pain as bad as it could be".
Clinical Outcome Measure - Back pain | 1-
  Decrease in Visual Analog Scale for Pain (VAS) for back by 3/10 or more at 24 months from the pre-operative value. Patients rated their back pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score fo 10 representing "pain as bad as it could be".

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Martinelli, Study Director — Geistlich Pharma AG
Locations (3):
- Germany (3):
  - Universitätsklinikum Augsburg - Neurochirurgische Klinik und Poliklinik, Augsburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Magdeburg gGmbH, Magdeburg

IPD SHARING:
Plan to Share IPD: No